CLINICAL TRIAL: NCT07336355
Title: A Randomized, Single-Blinded, Sham-Controlled Study Evaluating the Efficacy and Safety of RELAY, a Device Enabling Both Local Anesthetic Delivery and Neuromodulation Following Knee Surgery: Single Arm Training Run-In Phase
Brief Title: Feasibility of an Analgesic Device Enabling Local Anesthetic Delivery and Neuromodulation After Knee Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Gate Science (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RELAY Knee Feasibility
Record Dates: First submitted 2026-01-10; First posted 2026-01-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Intervention Model Description: A series of participants all receiving active treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental Treatment (Experimental): RELAY catheter will be inserted under ultrasound guidance followed by a local anesthetic bolus injection. Within the recovery room, the stimulators will be connected to participants' phones and turned on. The catheters will be removed on postoperative day 7.
  Interventions: Device: Percutaneous peripheral nerve stimulation

INTERVENTIONS:
Device: Percutaneous peripheral nerve stimulation — Percutaneous peripheral nerve stimulation with a frequency between 1-250 Hz, a pulse duration of 1-200 µs, and a current of 0.001-10 mA (1-10,000 µA). If the same pattern holds for the RELAY device as for previously tested peripheral nerve stimulators, we will maximize frequency, minimize pulse duration, and have participants adjust the amplitude, as needed.
  Other Names: femoral neuromodulation

SUMMARY:
Postoperative pain remains undertreated with inadequate analgesic options. Opioids have well-known limitations for both individuals and society; single-injection and continuous peripheral nerve blocks provide intense analgesia but are limited in duration to 24-72 hours; and current neuromodulation options-with a duration measured in weeks and not hours-are prohibitively expensive and require an additional procedure. One possible solution is a device currently under investigation to treat postoperative pain. The RELAY system (Gate Science, Moultonborough, New Hampshire) is comprised of a basic catheter-over-needle device to allow administration of a single-injection of local anesthetic via the needle (or catheter) followed by a perineural local anesthetic infusion via the remaining catheter (when desired). Subsequent to the local anesthetic administration, instead of removing the catheter as with all previous continuous peripheral nerve block equipment, electric current may be delivered via the same catheter and an integrated pulse generator for up to 28 days. This is potentially revolutionary because it would allow an anesthesiologist to deliver (1) a single-injection peripheral nerve block; (2) a continuous peripheral nerve block; and (3) neuromodulation using a single device that can theoretically be placed in the same amount of time required for a single-injection peripheral nerve block. Instead of providing fewer than 24 hours of postoperative analgesia, up to 28 days of pain control could be delivered without disruption of existing practice patterns. The ultimate objective of the proposed investigation is to prepare for a randomized clinical trial investigating the use of the RELAY device to provide postoperative analgesia.

This feasibility study will be a series of participants all receiving both local anesthetic and electric current via a single device (RELAY, Gate Science, Moultonborough, New Hampshire). The purpose will be to optimize the insertion approach and stimulation administration during the first 7 days following foot and shoulder surgery as well as training the clinical investigators.

DETAILED DESCRIPTION:
Specific Aim: To determine the feasibility and optimize the protocol for the RELAY device following foot and shoulder surgery to prepare for the subsequent randomized, controlled pilot study.

For individuals of childbearing potential, a sample of urine will be collected before any study interventions to confirm a non-pregnant state (this is standard procedure for all surgical patients). The RELAY device combines a catheter-over-needle to permit ultrasound-guided percutaneous insertion with the tip adjacent to a peripheral nerve or plexus, followed by needle removal which leaves the catheter in situ to deliver a bolus of local anesthetic (if desired) and subsequent perineural local anesthetic infusion (if desired). The catheter also has 3 integrated electrodes to enable neuromodulation using the integrated pulse generator and battery.

Participants will have standard external monitors placed and oxygen delivered by facemask or nasal cannula. The peripheral nerve block site(s) will be cleansed with chlorhexidine gluconate and isopropyl alcohol. Intravenous sedation/analgesia with midazolam and/or fentanyl will be titrated for patient comfort as is standard for peripheral nerve block administration. For knee surgery, the saphenous branch of the femoral nerve will be treated in the adductor canal with the long-acting peripheral nerve block (standard of care), and the experimental lead will be inserted by the femoral nerve near the inguinal crease. The target nerve(s) will be visualized with ultrasound using a transverse cross-sectional (short axis) view and a skin wheal of local anesthetic will be raised inferior to the transducer to anesthetize the skin and then the track towards the target. The RELAY with the integrated needle will be inserted adjacent to the femoral nerve with an in-plane approach. Dextrose 5% in water (1-20 mL) will be injected via the needle to open a space around the target nerve(s), the catheter advanced, and the needle subsequently withdrawn.

Electrical current will be introduced with increasing intensity via each of the anode electrodes to optimize participant's perceived stimulation (control provided by the Gate Keeper app from an investigator's phone or tablet). Accurate lead placement will be confirmed with subject reports of comfortable sensations over the thigh without eliciting muscle contractions. The minimum threshold and maximum comfortable amplitudes will be determined along with the optimal frequency, pulse duration, and anode/cathode. Starting from the lowest possible current the investigators increase the current until the participant states that they feel a "buzzing" sensation (some describe it as a "comfortable massage"). That is the minimal sensed current. The investigators then continue increasing with the instructions to let us know when it starts to be less comfortable-and to stop us before it hurts. That is the maximum comfortable current. The stimulator will be then set to deliver the minimum threshold amplitude and turned off for surgery. The pulse generator of the RELAY has a frequency between 1-250 Hz, a pulse duration of 1-200 µs, and a current of 0.001-10 milliamperes (1-10,000 milliamperes). The investigators will maximize frequency, minimize pulse duration, and have participants adjust the amplitude following surgery, as needed.

Local anesthetic (10 mL of lidocaine 2% with epinephrine) will be injected with negative aspiration every 3 mL and resulting sensory block confirmed to ensure accurate catheter tip placement. Following block confirmation (sensory deficits in the expected nerve distributions), the RELAY will be affixed with both surgical adhesive (2-Octyl 2-cyanoacrylate) at the entry site and a chlorohexidine-impregnated occlusive dressing [research specific]. Subsequently, 10 mL of bupivacaine 0.5% with epinephrine will be injected negative aspiration every 3 mL along with a supplemental single-injection saphenous nerve block.

Intraoperatively, surgeons will be permitted to infiltrate the surgical area with long-acting local anesthetic as their common practice dictates.

Postoperatively, the stimulators will be connected to participants' phones and turned on. After 7 days, participants themselves or their caretaker will remove the occlusive dressing and withdraw the catheter (and integrated electrodes) with gentle traction and counter-clockwise rotation at home. The devices are single-use and disposable.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants of at least 18 years of age
2. Undergoing a rotator cuff repair, total shoulder arthroplasty, ankle arthroplasty/arthrodesis, or foot surgery anticipated to result in moderate-to-severe pain for at least one week
3. Planned single-injection peripheral nerve block(s)
4. An Android or Apple smart phone able to download the Gate Keeper controller app

Exclusion Criteria:

1. Chronic opioid or tramadol use (daily within prior 2 weeks and duration > 4 weeks)
2. Neuro-muscular deficit of the surgical limb
3. Compromised immune system based on medical history (e.g., immunosuppressive therapies such as chemotherapy, radiation, sepsis, infection), or other conditions that places the subject at increased risk of infection
4. Implanted spinal cord stimulator, cardiac pacemaker/defibrillator, deep brain stimulator, or other implantable neurostimulator whose stimulus current pathway may overlap
5. History of bleeding disorder
6. Antiplatelet or anticoagulation therapies other than aspirin
7. Allergy to skin-contact materials (occlusive dressings, bandages, tape etc.)
8. Incarceration
9. Pregnancy
10. Moderate pain (NRS > 3) in an anatomic location other than the surgical site
11. Anxiety disorder
12. History of substance misuse
13. Inability to communicate with the investigators
14. Inability to contact the investigators during the treatment period, and vice versa (e.g., lack of telephone access)
15. Allergy to amide local anesthetics
16. Morbid obesity (body mass index > 40 kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Average Daily Pain Intensity 1st Week [Time Frame: Days 1-4 and 7] | Days 1-4 and 7
  The median of 5 daily "average" pain intensity scores for Days 1-4 and 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)

SECONDARY OUTCOMES:
Cumulative opioid use 1st week | The first 7 days following surgery
  The cumulative opioid use measured in oxycodone equivalents during the first 7 days following surgery
Brief Pain Inventory (Interference Sub Scale) Day 3 | Postoperative day 3
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale; (2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include solely the interference subscale with a minimum score of 0 (optimal outcome) and maximum score of 70 (worst possible outcome).
Brief Pain Inventory (Interference Sub Scale) Day 7 | Postoperative day 7
  The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale; (2) percentage of relief provided by pain treatments with one question [reported score is the percentage divided by 10 and then subtracted from 10: 0=complete relief,10=no relief] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include solely the interference subscale with a minimum score of 0 (optimal outcome) and maximum score of 70 (worst possible outcome).
Worst Daily Pain Intensity 1st Week | Days 1-4 and 7
  The median of 5 daily "worst" (maximum) pain intensity scores for Days 1-4 and 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Awakenings Due to Pain 1st Week | Collected on postoperative days 1, 2, 3, 4, and 7
  Cumulative number of nightly awakenings due to pain
Average Daily Pain Intensity Day 7 | Day 7
  The "average" pain intensity score on Day 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Worst (Maximum) Daily Pain Intensity Day 7 | Day 7
  The "worst" pain intensity score on Day 7 as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Opioid consumption Day 7 | Day 7
  The cumulative opioid use from the previous 24 hours measured in oxycodone equivalents as recorded on Day 7
Daily "Average" Pain Intensity | postoperative Days 1, 2, 3, 4, 7, 8 and 14
  The "average" pain intensity score on each postoperative day as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Daily "Worst" Pain Intensity | postoperative Days 1, 2, 3, 4, 7, 8 and 14
  The "worst" pain intensity score on each postoperative day as measured with the Numeric Rating Scale (0 minimum=best; 10 maximum=worst)
Daily Opioid Consumption | postoperative Days 1, 2, 3, 4, 7, 8 and 14
  The cumulative opioid use from the previous 24 hours measured in oxycodone equivalents as recorded on Days 1-4, 7, 8, and 14

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
A data sharing agreement with the university will be required
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately without a set duration limit